CLINICAL TRIAL: NCT00935545
Title: A Phase I Study of Peptide Vaccination With Tumor Associated Antigens Mixed With Montanide ISA-51VG in Pediatric Patients With Recurrent or Refractory Central Nervous System Tumors
Brief Title: Study of Peptide Vaccination With Tumor Associated Antigens Mixed With Montanide in Patients With CNS Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 08-1017
Record Dates: First submitted 2009-07-07; First posted 2009-07-09 (Estimated); Last update posted 2016-01-26 (Estimated); Status verified 2016-01

CONDITIONS: Tumors, Central Nervous System
Keywords: Brain Tumors; High Grade; CNS
MeSH Terms: conditions — Central Nervous System Neoplasms; Brain Neoplasms | interventions — Monatide (IMS 3015)

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Open Label (Experimental)
  Interventions: Biological: Montanide

INTERVENTIONS:
Biological: Montanide — Montanide is an oil-based immunoadjuvant similar to Incomplete Freund´s Adjuvant, which is commonly used in combination with peptide vaccines. Although its precise mode of action is not known, it acts to enhance the immune response to vaccination. It has a depot effect that depending on the type of emulsion will release the antigen slowly from the injection site.
  Other Names: Montanide ISA-51 VG

SUMMARY:
This is an open-label, single arm study evaluating a multi-peptide (tumor-associated antigens)/Montanide vaccine in patients < 21 years of age with recurrent or refractory CNS tumors. The study primarily evaluates the safety of this regimen. Secondarily, immunogenicity and anti-tumor effects will be assessed.

The primary aim is to evaluate the safety of subcutaneous injections of tumor associated antigens (TAA) mixed with Montanide ISA-51VG in patients with recurrent or refractory brain tumors.

The secondary aims are to evaluate cellular immune responses induced in patients after subcutaneous injection of TAA mixed with Montanide ISA-51VG and to document tumor response in patients with measurable disease or time to progression in patients without measurable disease following subcutaneous injection of TAA mixed with Montanide ISA-51VG.

ELIGIBILITY:
Inclusion Criteria

1. Patients with primary central nervous system tumors recurrent or refractory to standard therapy. Patients with recurrent tumors other than refractory anaplastic astrocytoma, glioblastoma multiforme or medulloblastoma must have failed all available second line therapies considered to be standard of care prior to inclusion in this study.
2. Patients with tumor histologies which have previously been shown to express at least one of the tumor associated antigens (TRP2, gp100, EphA2 or Her2) are eligible. Patients whose tumors are shown to express at least one of these antigens are also eligible.
3. Patients must be HLA A*0201 positive.
4. Age < 21 years
5. Patients must weigh > 15kg due to the amount of blood required for immune function studies.
6. Lansky performance status or Karnofsky performance status > 50. Patients who are unable to walk because of paralysis but who are up in a wheelchair, will be considered ambulatory for the purpose of assessing the performance score.
7. Adequate organ function:

   Hematologic: WBC > 1000/mm3 Absolute lymphocyte count > 500 Hemoglobin > 9 gm/dl (may be transfused to achieve adequate hemoglobin level) Platelet count > 50,000/mm3 INR and PTT < 1.5 x the upper limit of normal

   Hepatic: AST/ALT < 2 x the upper limit of institutional normal Total bilirubin < 1.5 x the upper limit of institutional normal

   Renal: Serum creatinine < upper limit of normal for the patient's age
8. Life expectancy > 3 months
9. Patients must have fully recovered from previous surgery, chemotherapy, radiotherapy and biologic therapy. No chemotherapy, radiation therapy or immunotherapy within 4 weeks prior to the first dose of study agent (6 weeks for nitrosureas)
10. Measurable disease is not required.
11. Informed consent must be signed by the patient or legal representative.

Exclusion Criteria

1. Serious illness, eg, uncontrolled infections requiring antibiotics.
2. History of immunodeficiency disease (such as HIV) or autoimmune disease except vitiligo.
3. Concomitant treatment with systemic corticosteroids greater than physiologic doses. Topical (but not at the proposed vaccination site) or inhalational steroids are permitted.
4. Participation in any other clinical trial involving another investigational agent within 4 weeks prior the first dose of study agent.
5. Pregnant or lactating women are not permitted.
6. Women of child-bearing potential not using medically acceptable means of contraception.

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 15 (Actual)
Dates: Start 2009-07; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
The primary aim is to evaluate the safety of subcutaneous injections of tumor associated antigens (TAA) mixed with Montanide ISA-51VG in patients with recurrent or refractory brain tumors. | 2-4 weeks

SECONDARY OUTCOMES:
Evaluate cellular immune responses induced in pts after injection of TAA mixed with Montanide and document tumor response in pts w/ measurable disease or time to progression in pts without measurable disease following injection of TAA mixed w/ Montanide. | 2-4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Sharon Gardner, MD, Principal Investigator — NYU Langone Medical Center
Locations (1):
- NYU Langone Medical Center, New York, New York, United States